CLINICAL TRIAL: NCT04838574
Title: Post-Chikungunya Rheumatism - Rheumatology Follow-up of Patients After 15 Years
Acronym: ChikRhuma15
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/03
Record Dates: First submitted 2021-03-19; First posted 2021-04-09 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Chikungunya
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 15 years Follow-up group — Phone recruitment, screening interview and eligibility questionnaire. Patient inclusion during rheumatologic evaluation : questionnaire, examination and data collection in one of the 4 study hospital centers.

SUMMARY:
Reunion Island was struck by a severe Chikungunya outbreak in 2005-2006. Three hundred and seven Chikungunya patients were evaluated by 4 rheumatologists 2 months after the initial infection (RHUMATOCHIK study). Eighty-three percents still reported joint pain and 43% joint swelling in telephone interviews after 32 months (Bouquillard et al., 2018). The primary objective of the present study is to assess and classify precisely persistent Chi-related joint diseases after 15 years, in a second rheumatology examination.

DETAILED DESCRIPTION:
Reunion Island was struck in 2005-2006 by the most severe Chikungunya outbreak (seroprevalence 38% (Gérardin et al., 2013)) in a developed but previously non-immunized country, providing an unique opportunity for studying Chikungunya-related joint symptoms and their long-term evolution. In a previous study, the investigators demonstrated that at least 17/73 patients initially classified as Chikungunya-related inflammatory joint diseases after 40 months still suffered from inflammatory joint symptoms fullfilling validated classification criteria after 13 years (Guillot et al., 2020). However, in this monocentric study, the investigators did not consider the full spectrum of Chikungunya-related rheumatic diseases, the population was not fully representative and the sample size was not sufficient to perform statistical analyses nor identify poor prognosis markers. In the RHUMATOCHIK cohort study, 307 patients were evaluated by 4 rheumatologists 2 months after the infection, 83% and 43% reported persistent joint pain and joint swelling respectively after 32 months in potentially biased telephone interviews (Bouquillard et al., 2018).

In this context, the present study aims at performing a systematic clinical rheumatologic re-evaluation of the RHUMATOCHIK patients after 15 years, in order to precisely describe and classify the full spectrum of persistent Chikungunya-related joint diseases in a larger population.

After a telephone interview and screening questionnaire, these patients will be clinically re-evaluated by a second rheumatologist in a multicenter transversal follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously included in the RHUMATOCHIK study (N=307), or diagnosed as Chikungunya-related Rheumatoid Arthritis (N=21) after telephonic screening and given their oral consent
* Chikungunya infection (positive serology and/or evocative symptoms in the epidemic context)

Exclusion Criteria:

* Impossible informed consent (cognitive impairment,…).
* Lost-to-follow-up patients, refusal to participate. -Pre-existing chronic inflammatory rheumatic disease (prior to CHIKV infection)-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients previously included in the RHUMATOCHIK study, or diagnosed as Chikungunya-related Rheumatoid Arthritis in the Reunion Island.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-02-19 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Describe the phenotype of chronic post-Chikungunya rheumatological pictures persisting 15 years after the initial infection | Day 0
  The primary outcome is the distribution (%) of rheumatic disease types among the patients with persistent Chikungunya-related rheumatic symptoms after 15 years ie. the percentage of patients fullfilling validated classification criteria of inflammatory rheumatic diseases (Rheumatoid Arthritis (Aletaha et al., 2010), Spondyloarthritis (Dougados et al., 1991; Rudwaleit et al., 2011a), Psoriatic Arthritis (Taylor et al., 2006), RS3PE - or undifferentiated arthritis), or classified in other rheumatic diseases (osteoarthritis, tendinitis, capsulitis, carpal tunnel syndrome, radicular pain, crystal-induced arthritis (Neogi et al., 2015), fibromyalgia (Wolfe et al., 2011)) - at inclusion.

SECONDARY OUTCOMES:
To describe the phenotype of post-Chikungunya chronic rheumatological pictures that have resolved 15 years after the initial infection. | Day 0
  The distribution (%) of rheumatic disease types among the patients with no more Chikungunya-related rheumatic symptoms after 15 years.
To specify the time of onset in relation to the initial infection of rheumatological pictures initially attributed to Chikungunya. | Day 0
  The mean duration (months) of Chikungunya-related rheumatic diseases.
Timing of onset of rheumatologic symptomatology in relation to CHIKV infection | Day 0
  Date of infection, date of onset of rheumatologic symptoms, time between the two (months), average duration (months) of rheumatologic symptomatology attributed to CHIKV infection
Rheumatological pictures pre-existing the infection | Day 0
  Comparison of patients with persistent versus resolving Chikungunya-related rheumatic diseases after 15 years, in order to identify prognostic factors

CONTACTS AND LOCATIONS:
Locations (3):
- Reunion (3):
  - CHU La Réunion (Nord), Saint-Denis
  - CH Ouest Réunion, Saint-Paul
  - CHU La Réunion (Sud), Saint-Pierre

IPD SHARING:
Plan to Share IPD: No